CLINICAL TRIAL: NCT04214106
Title: Thiamine Administration and Prevalence of Delirium in the Intensive Care Unit: A Before-after Study
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Brian Fredman, Dr., Meir Medical Center
Other Study IDs: 0277-19-MMC
Record Dates: First submitted 2019-12-08; First posted 2020-01-02 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Thiamine group: group 1: ICU patients who did not receive IV thiamine
- Non-thiamine group: group 2: ICU patients who received IV thiamine,100-500 mg/day for at least one day
  Interventions: Drug: intravenous Thiamine

INTERVENTIONS:
Drug: intravenous Thiamine — patients who received Thiamine,100-500 mg/day for at least one day
  Groups: Non-thiamine group

SUMMARY:
Delirium is a very common condition among ICU-admitted patients, and its prevalence is estimated between 30-40%. Delirium is associated with increased morbidity and mortality and future cognitive decline, along with increased ventilation-dependency and other complications.

There are multiple risk factors for delirium, including deficiencies of micronutrients. Thiamine deficiency is associated with specific neurological syndromes, including Wernicke and Korsakoff syndromes and Delirium Tremens. Several studies demonstrated significant thiamine deficiency among ICU-admitted patients (prevalence of 30-70%) without known risk factors, such as alcohol dependency. Thiamine deficiency may cause delirium in those patients.

Intravenous thiamine had been safely used for decades, for several indications. Lately, thiamine has been advocated for therapy in patients with septic shock, and its use in intensive care units has increased worldwide.

Since 2016, thiamine has been routinely administered in our intensive care unit. Considering the theoretical association between thiamine deficiency and ICU-related delirium, the investigators aim to investigate whether the routine use of thiamine has been associated with decreased prevalence of delirium among ICU patients when compared to the pre-routine thiamine administration era.

DETAILED DESCRIPTION:
Delirium is a very common condition among ICU-admitted patients, and its prevalence is estimated between 30-40%. Delirium is associated with increased morbidity and mortality and future cognitive decline, along with increased ventilation-dependency and other complications.

There are multiple risk factors for delirium, including deficiencies of micronutrients. Thiamine deficiency is associated with specific neurological syndromes, including Wernicke and Korsakoff syndromes and Delirium Tremens. Several studies demonstrated significant thiamine deficiency among ICU-admitted patients (prevalence of 30-70%) without known risk factors, such as alcohol dependency. Thiamine deficiency may cause delirium in those patients.

Intravenous thiamine had been safely used for decades, for several indications. Lately, thiamine has been advocated for therapy in patients with septic shock, and its use in intensive care units has increased worldwide.

Since 2016, thiamine has been routinely administered in our intensive care unit. Considering the theoretical association between thiamine deficiency and ICU-related delirium, the investigators aim to investigate whether the routine use of thiamine has been associated with decreased prevalence of delirium among ICU patients when compared to the pre-routine thiamine administration era.

Primary endpoint: Average delirium score during ICU-hospitalization before and after the routine intravenous thiamine administration.

Secondary endpoints: ICU and hospital admission times, duration of ventilation, need for tracheostomy, need for anti-delirium therapy and 28-day mortality.

Study design: Retrospective before-after interventional study. Inclusion criteria: All patients, aged 18-99, admitted to the intensive care unit in our medical facility between the years 2014-2018 (two years before and after intervention).

Exclusion criteria: Patients who were treated with thiamine prior to ICU admission, and patients who did not receive thiamine in the ICU.

Data collection: Data will be collected from the patients' electronic management file (iMD soft, Ofek and Chameleon software). Data collection will be anonymous.

Data: Age, gender, ICU and hospital admission times, duration of ventilation, 28-day mortality, need for tracheostomy. Need for anti-delirium therapy, cause for ICU admission, medical history, regular medication therapy, APACHE-2 score, SOFA score, lactate levels, need for inotropic or vasopressor support, need for physical restraints, need for renal replacement therapy, use of medication which may increase risk for delirium, RASS score.

Cohort size: 1000 patients overall, 500 in each study group (before and after intervention).

ELIGIBILITY:
Inclusion Criteria:

* All patients, aged 18-99, admitted to the intensive care unit in our medical facility between the years 2014-2018 (two years before and after intervention).

Exclusion Criteria:

* Patients who were treated with thiamine prior to ICU admission, and patients who did not receive thiamine in the ICU.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients, aged 18-99, admitted to the intensive care unit in our medical facility between the years 2014-2018 (two years before and after intervention).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Delirium score | Average RASS score during ICU-hospitalization, through study completion, an average of 1 year
  RASS score (Richmond agitation-sedation scale, from minus 5 to plus 4, desirable score 0)

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center Kfar Saba, Kfar Saba, Israel